CLINICAL TRIAL: NCT01695941
Title: A Phase I Study of MLN8237 in Combination With Bortezomib and Rituximab in Relapsed and Refractory Mantle Cell and Low Grade Non-Hodgkin Lymphoma
Brief Title: Alisertib, Bortezomib, and Rituximab in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma or B-cell Low Grade Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01712; NCI-2012-01712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S12-02028; CDR0000740877; P9086; 9086 (Other: Montefiore Medical Center - Moses Campus); 9086 (Other: CTEP); P30CA013330 (NIH)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Mantle-Cell | interventions — MLN 8237; Bortezomib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (alisertib, bortezomib, and rituximab) (Experimental): Patients receive alisertib PO BID on days 1-7; bortezomib SC on days 1, 8, and 15; and rituximab IV on day 1. Treatment repeats every 28 days* in the absence of disease progression or unacceptable toxicity.
  Note: *After 8 courses, treatment with rituximab repeats once every 3 courses (12 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN 8237; MLN-8237; MLN8237
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase I trial studies the side effects and best dose of alisertib and bortezomib when given together with rituximab in treating patients with mantle cell lymphoma or B-cell low grade non-Hodgkin lymphoma that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Alisertib and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Giving alisertib and bortezomib together with rituximab may be a better treatment for relapsed or refractory mantle cell lymphoma or B-cell low grade non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of alisertib (MLN8237) and bortezomib when combined with rituximab in patients with relapsed/refractory mantle cell and B-cell low grade non-Hodgkin lymphoma.

SECONDARY OBJECTIVES:

I. To describe the rate of overall response (complete response and partial response) for patients with relapsed/refractory mantle cell and B-cell low grade non-Hodgkin lymphoma treated with the combination of MLN8237 plus bortezomib and rituximab.

TRANSLATIONAL OBJECTIVES:

I. To evaluate the clinical significance of Aurora A over-expression and the proliferative index in initial tumor biopsy specimens from patients with relapsed/refractory mantle cell and B-cell low grade non-Hodgkin lymphoma treated with the combination of MLN8237 plus bortezomib and rituximab.

II. To evaluate and compare in paired biopsy specimens pre-treatment and on day 8: apoptosis and G2M arrest, and the expression level of cell cycle related proteins including: cyclin D1, p53, BIM-1, p27, p21, noxa, puma and survivin.

OUTLINE: This is a dose-escalation study of alisertib and bortezomib.

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7; bortezomib subcutaneously (SC) on days 1, 8, and 15; and rituximab intravenously (IV) on day 1. Treatment repeats every 28 days* in the absence of disease progression or unacceptable toxicity.

Note: *After 8 courses, treatment with rituximab repeats once every 3 courses (12 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed or refractory mantle cell lymphoma or low grade B-cell non-Hodgkin lymphoma (NHL); patients with evidence of transformation to a high grade histology will not be eligible
* Measurable or evaluable disease, as defined in 2008 Revised Response Criteria for Malignant Lymphoma; baseline scans used for measurement should be obtained within 30 days of registration, and baseline bone marrow biopsy and/or aspiration should be obtained with 90 days of registration
* Patients may have received one or more lines of prior chemotherapy with/without rituximab (including high dose therapy plus stem cell transplant which is counted as one regimen); prior bortezomib is allowed; patients must not have received bortezomib in the past 6 months
* Patients with human immunodeficiency virus (HIV) who are not receiving cytochrome p450 inhibitors, and who have a minimum of 300+ CD4+ cells/mm^3, an undetectable viral load, and no history of acquired immune deficiency syndrome (AIDS) indicator conditions
* Patients must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL (obtained within 30 days of registration)
* Absolute neutrophil count >= 1,500/mcL (obtained within 30 days of registration)
* Platelets >= 75,000/mcL or >= 50,000/mcL with documented bone marrow involvement (obtained within 30 days of registration)
* Total bilirubin within normal institutional limits (may be elevated if direct bilirubin normal) (obtained within 30 days of registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 X institutional upper limit of normal (obtained within 30 days of registration)
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (obtained within 30 days of registration)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MLN8237 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C, 3 weeks for rituximab) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN8237, bortezomib or rituximab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen, or any conditions that could result in excessive toxicity associated with the benzodiazepine-like effects of MLN8237
* Inability to swallow oral medication or to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration or any condition that would modify small bowel absorption of oral medications, including malabsorption, or resection of pancreas or upper bowel
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MLN8237
* HIV-positive patients on combination antiretroviral therapy which include cytochrome p450 inhibitors are ineligible; patients with CD4 counts less than 300 CD4+ cells/mm^3 and or a high viral load are ineligible
* Grade 2 or greater neuropathy
* The following agents are not permitted while patients are taking MLN8237, and should be discontinued at prior to registration if patients are taking them:

  * Patients must stop using the proton pump inhibitor (PPI) for at least 4 days prior to the first dose of MLN8237; administration of PPI while on study is not permitted
  * Histamine-2 (H2) receptor antagonists are not permitted from the day prior through to the end of MLN8237 dosing, except as required for premedication for rituximab; constant dosing of H2 blockers is not permitted
  * Antacid preparations are not permitted for 2 hours before or 2 hours after administration of MLN8237
  * Administration of pancreatic enzymes is not permitted at any time while on study
  * Co-administration of enzyme-inducing antiepileptic drugs, rifampin, rifabutin, rifapentine or St. John's wort is not permitted
  * Concurrent bisphosphonate therapy is allowed if it was started before study entry and is maintained at recommended dosing intervals; if bisphosphonate therapy is initiated after study entry, bone lesions will not be considered evaluable for disease response
  * Patients must be willing not drive, operate dangerous tools or machinery, or engage in any other potentially hazardous activity that requires full alertness and coordination if they experience excessive sedation; if a patient experiences excessive sedation believed to be related to MLN8237, treatment with MLN8237 should be interrupted
  * Patients must be willing to limit alcohol consumption to no more than 1 standard unit of alcohol (12 oz beer [350 mL], 1.5 oz [45 mL] of 80-proof alcohol, or one 6-oz [175 mL] glass of wine) per day during the study and for 30 days from the last dose of MLN8237; minimize the use of agents with central nervous system (CNS) effects
  * Benzodiazepine use is discouraged but not prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of alisertib when combined with bortezomib and rituximab, defined as the highest dose level at which < 33% of the dose cohort experience a dose limiting toxicity (DLT) | 21 days
  Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicities will be described by intensity at each dose level.
Recommended phase II dose of bortezomib when combined with alisertib and rituximab, defined as the highest dose level at which < 33% of the dose cohort experience a dose limiting toxicity (DLT) | 21 days
  Graded using the NCI CTCAE version 5.0. Toxicities will be described by intensity at each dose level.

SECONDARY OUTCOMES:
Overall response rate (ORR) (complete response and partial response) | Up to 30 days post-treatment
  ORR will be summarized descriptively.
Progression free survival (PFS) | From time of study entry to the first documentation of tumor progression or death due to any cause, whichever comes first, assessed up to 30 days post-treatment
  Kaplan-Meier methodology will be used to summarize estimate median PFS for patients in all treatment groups.
Duration of response (DOR) | From time of documentation of a response to treatment to the first documentation of documentation of tumor progression or death due to any cause whichever comes first, assessed up to 30 days post-treatment
  Kaplan-Meier methodology will be used to summarize estimate median DOR for patients in all treatment groups.
Overall survival | From time of randomization to the date of death due to any cause, assessed up to 30 days post-treatment

OTHER OUTCOMES:
Aurora A expression measured from patient biopsy specimens | Up to day 8 (course 1)
  Statistical techniques such as T-tests for bivariate analyses and logistic regression modeling for multivariable analyses will be applied to assess the association between initial Aurora A expression measured from patient biopsy specimens with response to therapy and other clinical outcomes. In patients who consent to biopsy, findings will be reported descriptively since these analyses will be viewed as exploratory in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Diefenbach, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (4):
- United States (4):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania